CLINICAL TRIAL: NCT04017624
Title: A Mobile Fresh Produce Market Intervention to Reduce Food Insecurity and Health Care Utilization Among Primary Care Patients in a Medicaid Accountable Care Organization: Randomized Pilot Study
Brief Title: Fresh Truck Pilot to Reduce Food Insecurity in a Medicaid ACO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID-19 pandemic impacted study methods. Therefore, the study team opted not to conduct this study as written. The study never started and no participants were enrolled.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38756
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Food Insecurity
Keywords: Mobile produce market; Boston Accountable Care Organization (BACO); Medicaid ACO; Accountable Care Organization; ACO; Social determinants of health; THRIVE; Healthcare utilization; Cost of care; Fruit and vegetable consumption
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh Truck with stipend (Experimental): Referral to Fresh Truck mobile market
  Interventions: Other: Fresh Truck with stipend
- THRIVE-Basic (Active Comparator): Screening-and-referral usual care model
  Interventions: Other: THRIVE screening and referral

INTERVENTIONS:
Other: Fresh Truck with stipend — Linkage to Community Partner Organization
  Investigators will partner with a community organization, Fresh Truck, that deploys mobile fresh produce trucks throughout Boston neighborhoods. Participants randomized to the intervention arm will receive a monthly stipend of $80 to purchase fresh produce available at any Fresh Truck mobile market location.
  Arms: Fresh Truck with stipend
Other: THRIVE screening and referral — The THRIVE screening tool includes questions to identify eight potentially unmet health-related social needs associated with health outcomes and healthcare utilization: housing and food insecurity, inability to afford medications, need for transportation, trouble paying for heat and electricity, need for employment or education, and difficulty taking care of children or other family members. The survey is written at a 3rd grade reading level, is available in multiple languages, and requires less than five minutes to complete. The paper screener consists of two parts: part one screens patients for health-related social needs in the eight domains. Part two asks patients to indicate the resources they want help accessing across the eight domains. Patients who request resources in one or more domains receive paper guides that describe available hospital and community resources to address the specific domain(s) indicated.
  Other Names: THRIVE-Basic
  Arms: THRIVE-Basic

SUMMARY:
This research is a randomized pilot study of an intervention to address food insecurity among intermediate risk Boston Accountable Care Organization (BACO) members receiving primary care at Boston Medical Center (BMC).

The investigators propose a parallel group, randomized pilot study among intermediate risk Medicaid ACO patients at BMC who have experienced food insecurity in the past 12 months, with a total enrollment of 120 participants (N=120). Half of the pilot study participants (n=60) will receive usual care: tailored printed paper referral guides to address health-related social needs, including resources for food insecurity (via the Health System's THRIVE Screening & Referral Program) and referrals to Boston Medical Center's Preventative Food Pantry. The other half (n=60) will receive access to a mobile fresh produce market and a monthly stipend to purchase items available on the mobile food trucks.

This pilot study will partner with Fresh Truck, a Boston-based 501(c)(3) organization that deploys mobile fresh produce trucks throughout Boston neighborhoods. Fresh Truck recently launched a new system, called 'Fresh Connect,' which addresses affordability as a barrier to healthy eating. 'Fresh Connect' enables healthcare systems to pay for fresh produce purchased by their patients from the Fresh Truck mobile markets.

The study protocol comprises three steps:

* Risk stratification before consent process to determine if the patient, at baseline, is within the top 3-20% of cost and utilization among BACO members. (This process is part of usual care operations in the Health System for ACO members).
* Of BACO patients identified as intermediate risk, patients will be screened for proximity to Fresh Truck mobile markets (zip code is among current Fresh Truck service area), nutritional need (food insecurity identified in the last 12 months), and not documented as housing insecure.
* Half the pilot study population will receive access to a mobile fresh food market intervention, Fresh Truck, and a stipend to purchase fresh produce aboard the trucks. The other half will receive usual care.

Pilot study participation is 6 months and will include collection and measurement of data from the following sources: baseline interview; final (6-months post-enrollment) interview, electronic medical records (EMR), BMC Clinical Data Warehouse (BMC CDW), and BMC HealthNet Plan (BMCHP) claims.

ELIGIBILITY:
Inclusion Criteria:

* Be within the 3rd to 20th percentile for healthcare utilization and cost among BACO membership at the time of enrollment into the pilot study
* Zip code that is in one of Fresh Truck's current services areas
* Documented as experiencing food insecurity in the previous 12 months
* Attend a primary care or ambulatory visit at BMC's primary care suites

Exclusion Criteria:

* Documentation of housing insecurity
* Receiving services from the BACO complex care management program

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in reported food insecurity based on the United States Department of Agriculture (USDA) food insecurity module | Baseline, 6 months
  The 6-item USDA food insecurity 30-day lookback module will be collected via interview at baseline and at 6 months

SECONDARY OUTCOMES:
Change in reported fruit and vegetable consumption | Baseline, 6 months
  A validated Fruit and Vegetable Consumption measure will be collected via interview at baseline and at 6 months
Change in food insecurity status based on THRIVE Screener | Baseline, 12 months
  Measured by the 2 questions relating to food insecurity in the BMC Health System THRIVE Screener
Total number of all-cause emergency department (ED) visits | Baseline, 6 months, 12 months
  Collected via BMC HealthNet Plan claims data
Total number of all-cause inpatient discharges | Baseline, 6 months, 12 months
  Collected via BMC HealthNet Plan claims data
Total patient-level cost of care | Baseline, 6 months, 12 months
  BMC HealthNet Plan claims data will be used to determine total cost of care

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverstein, MD MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No